CLINICAL TRIAL: NCT06092840
Title: Effect of a Thermogenic Composition on Healthy Adult Women and Men in a 12-week Weight Management Study
Brief Title: Effect of Transform Burn on Weight Loss
Acronym: Transform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4Life Research, LLC (Industry)
Collaborators: Brigham Young University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSC-009-01
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transform Burn (Experimental): Participants were supplied with one bottle of study product (Transform Burn) for each visit, labeled with their participant number. They were required to take the product consisting of 4 capsules per day, taken on an empty stomach at least 30 minutes prior to eating each morning, 5 days on Monday through Friday. Product was taken at the beginning of each visit, except for Week 0 visit for a total of 12 weeks and bottles were returned at each visit.
  Interventions: Dietary Supplement: Transform Burn

INTERVENTIONS:
Dietary Supplement: Transform Burn — Study product Transform Burn contains dihydrocapsiate, red pepper (Capsicum annuum) fruit extract, citrus (Citrus spp) peel extract, coleus (Coleus forskholi) root extract, and african mango (Irvingia gabonensis) seed extract.
  Other Names: Active Treatment

SUMMARY:
This study was undertaken to explore the effects of a Thermogenic Composition (TC) composed of dihydrocapsiate, red pepper (Capsicum annuum) fruit extract, citrus (Citrus spp) peel extract, coleus (Coleus forskholi) root extract, and african mango (Irvingia gabonensis) seed extract to support body composition, weight management, and improve parameters related to energy, hunger, and satiety on healthy adult women and men over a 12-week interval.

ELIGIBILITY:
Inclusion Criteria:

* Individuals could participate who were at least 18 years old and not smokers.
* Not currently taking a dietary supplement or prescription for weight loss.
* Exercising volunteers were asked to maintain their regimen consistently throughout the course of the 12-week study and caffeine drinking volunteers maintained their caffeine intake consistently throughout the course of the 12-week study.

Exclusion Criteria:

* Participants were not allowed to participate if they were pregnant or planning to become pregnant in the following 12 weeks, or lactating.
* Individuals were not allowed to participate if they were taking any stimulant medications.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Satiety Score | 12 weeks
  Results obtained from a validated ten-point scale Visual Analog Scale (VAS). On a scale 1 - 10, with the lowest being 1 and the highest being 10.
Resting Metabolic Rate | 12 weeks
  Resting metabolic rate (RMR) was measured by MedGem by MicroLife Medical Home Solutions, participants were in quiet, thermo-neutral environment, in a seated position, resting in a comfortable or reclined position for 5-15 minutes prior to measurement, without caffeine, food or exercise for at least four hours, with mouth-piece and nose-clip on, making sure of a good seal around the mouth and nose, holding MedGem device with arm support (e. g., pillow or opposite hand).
Blood Pressures | 12 weeks
  Both systolic and diastolic pressures were measured using the Omron Intellisense digital blood pressure monitor, Model HEM-739. Participants were measured in a seated position, left arm rested on the chair (or table) so that the cuff was at the same level as the heart, returned the palm upward, remained still and not talk.
Heart Rates | 12 weeks
  Heart rates were measured using the Omron Intellisense digital blood pressure monitor, Model HEM-739. Participants were measured in a seated position, left arm rested on the chair (or table) so that the cuff was at the same level as the heart, returned the palm upward, remained still and not talk.
Glucose Levels | 12 weeks
  Glucose levels were measured by CardioChek Plus. Participants were measured in a seated position with the index finger cleaned with an alcohol wipe dry until dried, a sterile lancet was used to puncture the skin on the side of the fingertip, around 100 microliter of blood was collected. With the glucose test strip already inserted into the device, 35-40 microliter of blood was applied to the test strip window and results appeared in approximately two minutes after.
Cholesterol Levels | 12 weeks
  Cholesterol levels were measured by CardioChek Plus. Participants were measured in a seated position with the index finger cleaned with an alcohol wipe dry until dried, a sterile lancet was used to puncture the skin on the side of the fingertip, around 100 microliter of blood was collected.
Body Fat | 12 weeks
  Body fat were measured by a pre-calibrated Tanita BC-418 Body Composition Analyzer, participants were measured in a standing position with shoes and socks removed, without exercise for at least four hours prior to the measurement, on an empty bladder, with both arms held straight down, not touching sides, inner thighs not touching, and feet cleaned.
Body Weight | 12 weeks
  Body weights were measured by a pre-calibrated Tanita BC-418 Body Composition Analyzer, participants were measured in a standing position with shoes and socks removed, without exercise for at least four hours prior to the measurement, on an empty bladder, with both arms held straight down, not touching sides, inner thighs not touching, and feet cleaned.
Waist and Hip Ratio (WHR) | 12 weeks
  Waist and hip circumference measurements were measured according to the US National Health and Nutrition Examination Survey III protocol. Participants were measured in a standing position, waist measurement was made at the high point of the iliac crest, hip measurement was made at the maximum extension of the buttocks, tape was parallel to the floor and snug, but not compressing skin.

CONTACTS AND LOCATIONS:
Overall Officials: David Vollmer, PhD, Principal Investigator — 4LIFE
Locations (1):
- 4Life Research, Sandy City, Utah, United States

IPD SHARING:
Plan to Share IPD: No